CLINICAL TRIAL: NCT03328975
Title: An Evaluation of Blood Glucose Levels and Insulin Requirement After Subacromial Corticosteroid Injection in Insulin Dependent Diabetics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to withdraw study
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bryson Lesniak, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO17070506
Record Dates: First submitted 2017-09-17; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Injury; Insulin-dependent Diabetics
MeSH Terms: conditions — Shoulder Injuries | interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): Group 1 will receive an injection of 4mg of dexamethasone 4 mL of 1% lidocaine.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Group 2 will receive an injection of 5 mL of 1% lidocaine (placebo).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — The overall purpose of this study is to evaluate the effect of a corticosteroid shoulder injection on glucose levels in insulin-dependent diabetic men and women.
  Other Names: Corticosteroid
  Arms: Dexamethasone
Other: Placebo — the placebo group will not receive the corticosteroid medication in their injection to treat the inflammation and pain in their shoulder. Instead, they will receive an injection of 5 mL lidocaine only.
  Arms: Placebo

SUMMARY:
The overall purpose of this study is to evaluate the effect of a corticosteroid shoulder injection on glucose levels in insulin-dependent diabetic men and women.

ELIGIBILITY:
Inclusion Criteria

* Insulin-dependent diabetic
* Age 18+
* Shoulder pain for over 4 weeks duration that is uncontrolled with activity modification or nonsteroidal anti-inflammatory drugs
* Use of glucometer for blood sugar monitoring
* Well controlled blood glucose levels
* Hemoglobin A1c less than or equal to 7.5

Exclusion Criteria

* Previous corticosteroid injection within the past 6 months
* Active infection
* Pregnant or plan on becoming pregnant
* Previous adverse event with corticosteroid or lidocaine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Can diabetic patients maintain their blood glucose in a normal range after receiving a corticosteroid injection? | 4 weeks
  The main outcome variable in this study is to determine what effects, if any, a corticosteroid injection has on the ability of diabetic patients to maintain their blood glucose in a normal range. This will allow for better patient education when discussing the risks of corticosteroid injections and allow for improved post-injection care of patients.